CLINICAL TRIAL: NCT02955303
Title: The Feasibility of TECH: Tablet Enhancement of Cognition and Health, Cognitive Training Using Touchscreen Tablet Gaming Applications, for Healthy Older Adults - a Pilot Randomized Control Trial
Brief Title: The Feasibility of TECH: Tablet Enhancement of Cognition and Health for Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Zvi Buckman, Dr. Zvi Buckman, Assuta Hospital Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016009-2
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy Adults
Keywords: Cognitive training; Tablet computers
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TECH protocol (Experimental): Daily self-training using tablet apps facilitated by weekly group sessions. The self-training will take place independently at participants' home and will include mostly playing puzzle-apps to train different cognitive components. Participants will be requested to play (and log) various apps three to five times a week for 30-60 minutes each time, for a total of 15-20 training sessions. In addition they will use the tablets for a variety of everyday uses. The individual self-training will be accompanied by five weekly sessions (of 60-90 minutes) in a small group setting (5-6 participants) led by an experienced occupational therapist. For initial learning of the tablet's basic use, an individual session for each participant will take place.
  Interventions: Other: TECH: Tablet Enhancement of Cognition and Health

INTERVENTIONS:
Other: TECH: Tablet Enhancement of Cognition and Health — cognitive training using touchscreen tablet gaming applications

SUMMARY:
This study assess the feasibility of novel cognitive intervention utilizing tablet apps (TECH protocol: Tablet Enhancement of Cognition and Health) in terms of relevance, adherence, suitable challenges, training time etc. for healthy older adults. Older adults with normal cognition will be randomly allocated to the TECH protocol (experimental group) or the control group (no treatment). Assessments will be administered pre and post the 6-week TECH protocol by assessors blind to group allocation.

DETAILED DESCRIPTION:
A pre-post pilot study will be conducted. Participants will be referred to the study from 'Maccabi Healthcare Services' by family physicians and geriatric physician of 'Maccabi Healthcare Services Central District'. The majority of TECH protocol training will take place in the participants' home as self-practice. The assessment and weekly group meetings will take place at clinics of Maccabi Healthcare Services in the Central District. A Helsinki approval (#2016009) has already been obtained. Participants will receive information regarding the study and if eligible will sign a consent form, undergo the screening and then the pre-intervention assessments. Then they will receive the TECH protocol, and following the intervention a second assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and above.
* Without cognitive decline (score 26 points or above in MoCA).
* ) live independently in the community (as reported by the participants, regarding their independence in BADL and IADL, excluding motor difficulties which are not caused due to neurological conditions or lack of performance with no changes compared to the past.
* Have normal or corrected vision and hearing.
* Speak, write and read Hebrew.
* Able to understand and follow use of the touchscreen of a tablet after initial demonstration.

Exclusion Criteria:

* Experience severe depressive symptoms (10 points or more in The Geriatric Depression Scale).
* Are diagnosed with dementia, or other neurological or psychiatric condition (such as stroke, Parkinson's disease).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Feasibility information | 7 minutes
  Information regarding: Adherence - the percentage of session attendance out of the six weekly group sessions; Compliance - assessed by the total self-training hours a week, which was taken from participant's daily logs and iPad Screen time information. Satisfaction from the intervention was rated by the participants after completion of the TECH intervention.

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment | 10 minutes
  A cognitive screening tool with high sensitivity and specificity, aimed to distinguish individuals with MCI from healthy adults. The MoCA assesses eight cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
WebNeuro | 20 minutes
  A computerized web-based battery assessment of neurocognitive functioning. The battery will include seven subtests that examine three cognitive domains: memory (Memory recognition/verbal list-learning task), executive planning (Switching of attention test, Verbal interference test, Maze test, Go-no-go test), and attention (Digit span test, Continuous performance test).
The Tower of Hanoi (ToH) task | 10 minutes
  A commonly used goal-directed measure assessing problem-solving, and specifically, planning. The ToH consists of three bars and three to eight different-sized disks that can slide onto any bar. The objective of the task is to move an entire stack (organized in ascending order of size on one bar) to another bar while obeying two rules: Only one disk can be moved at a time and no disk may be placed on top of a smaller disk. The score of the task is the number of moves for achieving each level. A computerized version of the task will be used (http://vornlocher.de/tower).

OTHER OUTCOMES:
The 12-Item Short Form Health Survey (SF-12) | 8 minutes
  SF-12 includes 12 questions from the SF-36 Health Survey. The SF-36 is a widely used and investigated, and validated instrument for measuring quality of life. The SF-12 was developed using normative data for the SF-36 in the United States. The shorter version designed to reproduce the Physical and the Mental Components Summary scores.
  A greater score indicates better health measures.
General Self-Efficacy Scale | 8 minutes
  Designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. It consists 10 statements such as 'I can solve most problems if I invest the necessary effort'. Possible responses are scored 1-4 (1 - not at all true to 4 - exactly true), the total score range from 10 to 40. Higher scores represent higher levels of general selfefficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Buckman, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided